CLINICAL TRIAL: NCT07157488
Title: Dual Task Training With Vestibular Stimulation in Children With Diplegic Cerebral Palsy
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Lahore (Other)
Responsible Party: Principal Investigator, Aqsa Majeed, Dr. Aqsa Majeed, University of Lahore
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Anam Mujahid
Record Dates: First submitted 2025-08-27; First posted 2025-09-05 (Actual); Last update posted 2025-09-05 (Actual); Status verified 2025-08

CONDITIONS: Diplegic Cerebral Palsy
Keywords: Diplegic cerebral palsy; Dual task training; Vestibular stimulation
MeSH Terms: conditions — Cerebral Palsy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Conventional Physical Therapy With Dual Task Training (Active Comparator): Participants receive conventional physical therapy combined with dual task training.
  Warm-up (10 min): Trunk and lower extremity ROM exercises (Lee et al., 2021).
  Conventional PT (20 min): Wide leg squatting, hip flexion/extension, hip abduction/adduction, knee extension/flexion with ankle weights (Uysal et al., 2024).
  Dual Task Training (20 min): Balance activities (semi-tandem stance, tiptoe, heel stance, one-leg stance, line walking) combined with cognitive tasks (verbal fluency, simple math, memory recall, daily routine recall).
  Session Duration: 50 minutes, 3 times/week for 12 weeks.
  Interventions: Behavioral: Conventional Physical Therapy With Dual Task Training; Behavioral: Dual Task Training With Vestibular Stimulation
- Dual Task Training With Vestibular Stimulation (Experimental): Participants receive dual task training combined with vestibular stimulation exercises.
  Warm-up (10 min): Trunk and lower extremity ROM exercises (Lee et al., 2021).
  Dual Task Training (20 min): Same protocol as Arm 1 (balance + cognitive tasks).
  Vestibular Stimulation (20 min): Sliding activity on physio roll (10 repetitions) and vertical bouncing while seated on physio roll for 10 minutes (Parashar et al., 2017).
  Session Duration: 50 minutes, 3 times/week for 12 weeks.
  Interventions: Behavioral: Conventional Physical Therapy With Dual Task Training; Behavioral: Dual Task Training With Vestibular Stimulation

INTERVENTIONS:
Behavioral: Conventional Physical Therapy With Dual Task Training — Participants undergo a 50-minute session, 3 times/week for 12 weeks.
  Warm-up (10 min): Trunk and lower extremity ROM exercises (Lee et al., 2021).
  Conventional PT (20 min): Wide leg squatting, hip flexion/extension, hip abduction/adduction, knee extension/flexion with ankle weights (Uysal et al., 2024).
  Dual Task Training (20 min): Balance activities (semi-tandem stance, tiptoe, heel stance, one-leg stance, line walking) with cognitive activities (verbal fluency, simple math, memory recall, daily routine recall).
Behavioral: Dual Task Training With Vestibular Stimulation — Participants undergo a 50-minute session, 3 times/week for 12 weeks.
  Warm-up (10 min): Trunk and lower extremity ROM exercises (Lee et al., 2021).
  Dual Task Training (20 min): Same as Intervention 1 (balance + cognitive tasks).
  Vestibular Stimulation (20 min): Sliding activity on physio roll (10 repetitions) and vertical bouncing on physio roll for 10 minutes (Parashar et al., 2017).

SUMMARY:
Dual task training enhances gross motor function, reduce fatigue and minimize cognitive motor interference in children with diplegic cerebral palsy by promoting neuroplasticity and improving dual task processing. Vestibular stimulation improve balance triggering the vestibulospinal reflex, which play a key role in maintaining posture and reducing the risk of fall. Integrating dual task training with vestibular stimulation can provide a more holistic rehabilitation strategy by enhancing balance and posture stability through improved vestibular system activation, supporting motor and cognitive coordination by challenging the brain to handle tasks concurrently, and boosting functional mobility by mimicking everyday situations that require divided attention. This RCT evaluates its effectiveness in optimizing motor-cognitive integration, functional mobility and endurance compared to conventional motor training approaches.

ELIGIBILITY:
Inclusion Criteria:

- Diagnosis of diplegic cerebral palsy (confirmed by physician/therapist).

Age between 6-12 years.

Gross Motor Function Classification System (GMFCS) levels II-III.

Ability to walk with or without assistive devices.

Stable medical condition for the past 6 months.

Parental/guardian consent to participate.

Exclusion Criteria:

* History of recent orthopedic surgery (within the past 6 months).

Botulinum toxin injections within the past 6 months.

Severe uncontrolled epilepsy or other uncontrolled medical conditions.

Severe cognitive impairment preventing ability to follow instructions.

Significant visual, auditory, or vestibular disorders unrelated to cerebral palsy.

Participation in another interventional clinical study within the last 3 months.

Ages: 6 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 54 (Estimated)
Dates: Start 2025-09 (Estimated); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Gross Motor Function Measure (GMFM-88) | Baseline and at 12 weeks (post-intervention, within 1 week of completion)
  The GMFM-88 is a standardized observational instrument designed to measure changes in gross motor function in children with cerebral palsy. Scores range from 0-100, with higher scores indicating better gross motor performance.

IPD SHARING:
Plan to Share IPD: No